CLINICAL TRIAL: NCT01399710
Title: Measure of Performances of CT Colonography With Computer-Aided Detection (CAD) as Second Reader in Detecting Colorectal Lesion
Brief Title: Impact of Computer-Aided Detection (CAD) as Second Reader in CT Colonography
Acronym: CAD-IMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: im3D S.p.A. (Other)
Collaborators: Candiolo Cancer Institute - IRCCS (Other); Bicocca Universiy of Milano, Milan, Italy (Unknown); Fondazione Salvatore Maugeri (Other); Catholic University, Italy (Other); Valduce Hospital (Other); University of Turin, Italy (Other); University of Roma La Sapienza (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Nuovo Regina Margherita Hospital (Other); University of Pisa (Other); University of Florence (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Daniele Regge, Institute of Cancer Research and Treatment, Candiolo - Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAD COLON 001
Record Dates: First submitted 2011-07-15; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Individuals With Suspected Colorectal Disease
Keywords: colorectal cancer; CT colonography; CAD
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Colonography, Computed Tomographic; Diagnosis, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: CT colonography — Participants were placed on a CT table and a small flexible rectal catheter was positioned. N-butyl-scopolamine was administered intravenously if this was common practice in the participating center. Immediately before scanning, pneumocolon was obtained through insufflation of room air or carbon dioxide, either manually by means of a balloon pump or with an automatic device, until maximum tolerance was reached. CT colonography was performed with the participant in supine and prone positions with the following scanning protocol: 120 kilovolt peak (kVp), 50 or fewer effective mA per second, and a section thickness not greater than 1.25 mm.
Procedure: colonoscopy — Colonoscopy was performed at least 3 hours after CT colonography. The endoscope was advanced to the cecum and the entire length of the bowel was examined during endoscope withdrawal. The endoscopist was initially blinded to the result of CT colonography; at the end of each bowel segment evaluation, CT colonography results for that segment were disclosed (segmental unblinding). If a lesion measuring 6 mm or larger was detected at CT colonography but not at colonoscopy, the segment was reexamined to resolve the discrepancy
Device: CT Colonography with computer assisted diagnosis (CAD),CADCOLON -im3D SpA., Torino Italy — Each CT colonography study was read in two phases. In the first phase the radiologist interpreted the examination without activating the CAD algorithm. This phase of reporting was defined as unassisted reading. Then the radiologist activated the CAD algorithm which pinpointed a series of colorectal lesion-like structures (i.e. lesion candidates) on both the prone and supine acquisition. All lesion candidates were examined. The second phase of reporting was defined as CAD-assisted reading.

SUMMARY:
RATIONALE: CT colonography accurately detects large polyps and masses. However, the test is less accurate in identifying lesions between 6 and 9 mm.Use of computer-aided detection (CAD) has shown promising results in providing uniform accuracy and improving CT colonography sensitivity.

PURPOSE:This clinical trial compared the performance of CT colonography with unassisted and CAD-assisted reading in detecting patients with colorectal lesions.

DETAILED DESCRIPTION:
Design: multicenter, cross-sectional study. Each participant underwent CT colonography and colonoscopy on the same day. Expert readers interpreted CT colonography unassisted and then reviewed all colorectal lesion-like structures pinpointed by the CAD algorithm.

ELIGIBILITY:
Inclusion Criteria:

- clinical indication to undergo colonoscopy either for symptoms, or participating a surveillance program or a CRC screening

Exclusion Criteria:

* clinical diagnosis of familial adenomatous polyposis or hereditary nonpolyposis CRC syndrome
* inflammatory bowel disease
* celiac disease
* evidence of increased risk of harm from colonoscopy
* psychological or physical conditions that contraindicated colonoscopy or CT Colonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CT colonography with unassisted and CAD-assisted reading in detecting individuals with lesions 6 to 9 mm
Specificity of CT colonography with unassisted and CAD-assisted reading in detecting individuals with no clinical relevant lesions

SECONDARY OUTCOMES:
Sensitivity of CT colonography with unassisted and CAD-assisted reading in detecting individuals with lesions 10 mm or larger
Sensitivity of CT colonography with unassisted and CAD-assisted reading in detecting lesions 6 mm or larger

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Regge, Principal Investigator — Institute Institute for Cancer Research and Treatment, Candiolo, Italy

REFERENCES:
- [Derived] Regge D, Della Monica P, Galatola G, Laudi C, Zambon A, Correale L, Asnaghi R, Barbaro B, Borghi C, Campanella D, Cassinis MC, Ferrari R, Ferraris A, Hassan C, Golfieri R, Iafrate F, Iussich G, Laghi A, Massara R, Neri E, Sali L, Venturini S, Gandini G. Efficacy of computer-aided detection as a second reader for 6-9-mm lesions at CT colonography: multicenter prospective trial. Radiology. 2013 Jan;266(1):168-76. doi: 10.1148/radiol.12120376. Epub 2012 Nov 14. PMID 23151831